CLINICAL TRIAL: NCT02250079
Title: Features and Differences Between Neonates Undergoing Body Bag With Polyethylene and Conventional Drying During Neonatal Adaptation in Maternal and Child Headquarters Hospital and the Victoria Hospital Engativá, Bogotá, 2013
Brief Title: Polyethylene Body Bags as an Alternative to Radiant Heat Lamp During the Neonatal Adaptation in Infants Older Than 29 Weeks
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universidad Nacional de Colombia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: polyethylene29
Record Dates: First submitted 2014-09-08; First posted 2014-09-26 (Estimated); Last update posted 2014-09-26 (Estimated); Status verified 2014-09

CONDITIONS: Neonatal Adaptation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Polyethilene body bag group (Experimental): The intervention group infants were provided the same care as control infants, but were dressed with the polyethylene body bag immediately after birth. The bag had an upper opening for the head and a seal at the bottom. The intervention group infants remained in the plastic bag for the first 10 minutes after birth. The same process was done in surgery room in case of cesarean. Umbilical prophylaxis, vitamin K1 application, initial physical examination and ocular prophylaxis are performed. The infants were swaddled in blankets provided by the mother, the head was covered with a hat, and the infants were placed either in an open crib or under a radiant warmer as necessary and available. The same process were done in surgery room in case of cesarean
  Interventions: Device: polyethylene plastic bag
- Conventional group (Active Comparator): ): Infants randomized to the control group received standard hospital care newborn. This included immediate drying, skin-to-skin contact, early and exclusive breast feeding, postponed bathing, bundling, and radiant warmer. While waiting for criteria cord clamping, the environment humidity and temperature and segment and rectal temperature of the newborn were measure. It was repeated at 1-5- 10-60 and 120 minutes. After clamping, the newborn were positioned in a radiant warmer, and completed the drying process. Umbilical prophylaxis, vitamin K1 application, initial physical examination and ocular prophylaxis are performed. The infants were swaddled in blankets provided by the mother, the head was covered with a hat, and the infants were placed either in an open crib or under a radiant warmer as necessary and available. The same process was done in surgery room in case of cesarean.
  Interventions: Device: Conventional treatment

INTERVENTIONS:
Device: polyethylene plastic bag — Inborn neonates with both a gestational age >29 weeks were randomized 1:1 to either a standard thermoregulation protocol or placement of a Poliethylene body bag since birth to 10 minutes after birth.
  Arms: Polyethilene body bag group
Device: Conventional treatment — Infants randomized to the control group received standard hospital care newborn. This included immediate drying, skin-to-skin contact, early and exclusive breast feeding, postponed bathing, bundling, and radiant warmer. While waiting for criteria cord clamping, the environment humidity and temperature and segment and rectal temperature of the newborn were measure. It was repeated at 1-5- 10-60 and 120 minutes. After clamping, the newborn were positioned in a radiant warmer, and completed the drying process. Umbilical prophylaxis, vitamin K1 application, initial physical examination and ocular prophylaxis are performed. The infants were swaddled in blankets provided by the mother, the head was covered with a hat, and the infants were placed either in an open crib or under a radiant warmer as necessary and available. The same process was done in surgery room in case of cesarean.
  Arms: Conventional group

SUMMARY:
INTRODUCTION: Hypothermia in the newborn causes morbid conditions. In developing countries in the basic technology for neonatal adaptation may not be available. Polyethylene bags may be an alternative to lamp radiant heat to prevent hypothermia OBJECTIVE: To characterize the differences between babies undergoing body bag with polyethylene or conventional drying during neonatal adaptation in the Hospital de la Victoria and Hospital de Engativá, Bogotá, Colombia, 2013.

MATERIALS AND METHODS: parallel-group randomized controlled trial. Groups: dried conventional (control) or polyethylene body bag (intervention). The procedure lasted 10 minutes, the bag body and / or radiant heat lamp was removed. Environment temperature and humidity, temperature in the body segments 1-5-10-60-120 minutes and APGAR was measured. Statistical Analysis: Descriptive bivariate statistical inference and calculated. Risk ratio (RR) and confidence intervals (CIs) were determined using contingency tables for risk analysis of the outcome. The study was approved by the hospital ethics committee of victory.

ELIGIBILITY:
Inclusion Criteria:

* Inborn neonates with both a gestational age >29 weeks

Exclusion Criteria:

* Abdominal wall defect, myelomeningocele, major congenital anomaly, or blistering skin disorder

Ages: 29 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2013-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Temperature | 10 minutes
  The Student's t test and U of Mann Whitney were used to compare temperature
Humidity | 10 minutes
  The Student's t test and U of Mann Whitney were used to compare relative humidity.

SECONDARY OUTCOMES:
Both, Hypothermia or Hyperthermia | 10 minutes
  Risk ratio (RR) and confidence intervals (CIs) were determined using contingency tables for risk analysis of hypothermia, hyperthermia and APGAR.

OTHER OUTCOMES:
Baseline Charasteristics | 10 minutes
  The baseline characteristics of each group were compared using descriptive statistics. The Student's t test and x2 were used to compare continuous and categorical variables, respectively. Fisher's exact test was used for events with low prevalence.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Victoria, Bogotá, Colombia